CLINICAL TRIAL: NCT06857747
Title: An Exploratory, Multicenter, Multi-cohort Phase II Clinical Trial of Disitamab Vedotin in Combination with Metronomic Chemotherapy in Advanced HER2-expressing Breast Cancer.
Brief Title: Disitamab Vedotin in Combination with Metronomic Chemotherapy in Advanced HER2-expressing Breast Cancer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: QIAO LI (Other)
Responsible Party: Sponsor-Investigator, QIAO LI, Clinial professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4532
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Vinorelbine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HER2-positive advanced breast cancer (Experimental): Patients will receive disitamab vedotin combining with metronomic chemotherapy in a 3-week treatment cycle.
  Interventions: Drug: Capecitabine; Drug: Vinorelbine; Drug: Etoposide
- HER2 2+/1+ expressed in IHC advanced breast cancer (Experimental): Patients will receive disitamab vedotin combining with metronomic chemotherapy in a 3-week treatment cycle.
  Interventions: Drug: Capecitabine; Drug: Vinorelbine; Drug: Etoposide

INTERVENTIONS:
Drug: Capecitabine — metronomic capecitabine, 500 mg, tid， po
Drug: Vinorelbine — metronomic vinorelbine, 40mg/d, TIW1, po
Drug: Etoposide — metronomic etoposide, 50mg/d, po

SUMMARY:
This study aims to explore the efficacy of Disitamab vedotin in combination with metronomic chemotherapy in advanced breast cancer. By integrating the rapid onset of action of Disitamab vedotin with the characteristics of metronomic chemotherapy, the study seeks to further improve patients' response rates and enhance their quality of life, building upon the extension of patient survival.

DETAILED DESCRIPTION:
Disitamab vedotin is a novel, cleavable antibody-drug conjugate (ADC) targeting HER2, with prior research indicating its efficacy in HER2-positive and low-expressing breast cancer. Patients with advanced breast cancer often have compromised general conditions, and some may have received conventional intensity chemotherapy, making further treatment challenging. Metronomic chemotherapy, characterized by lower drug doses, reduced intensity, continuous administration, and fewer adverse effects, offers the potential to improve quality of life and prolong survival for these patients. This study aims to explore the efficacy of disitamab vedotin in combination with metronomic chemotherapy in advanced breast cancer. By combining the rapid onset of action of disitamab vedotin with the characteristics of metronomic chemotherapy, the study seeks to not only extend patient survival but also enhance response rates and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign an informed consent form;
2. Male or female, aged ≥18 years;
3. Expected survival period ≥12 weeks;
4. Patients with histologically confirmed HER2-positive advanced breast cancer;
5. Measurable lesions as defined by RECIST v1.1 criteria;
6. Ability to provide tumor samples for HER2 testing from the primary or metastatic lesion:

   * HER2-positive definition: confirmed by immunohistochemistry (IHC) score of 3+ or 2+/fish+;
   * HER2 low expression definition: confirmed by IHC score of 2+/1+;

   Previous treatment requirements:
   * HER2 3+: previously received at least 1 line of treatment;
   * HER2 low HR+: progression after prior endocrine therapy and <3 lines of chemotherapy;
   * HER2 low HR-: <3 lines of chemotherapy in the past;
7. ECOG performance status score 0-1;
8. Adequate cardiac, bone marrow, liver, and renal function (according to the normal values of the research center):

   Hematologic criteria:
   * Hemoglobin (Hb) ≥ 100 g/L;
   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   * Platelet count (PLT) ≥ 100 × 10^9/L;

   Biochemical criteria:
   * For patients without liver metastases, ALT and AST ≤ 3 × ULN, serum total bilirubin ≤ 1.5 × ULN;
   * For patients with liver metastases, ALT and AST ≤ 5 × ULN, serum total bilirubin ≤ 3 × ULN;
   * Serum creatinine (Cr) ≤ 1.5 ULN or estimated creatinine clearance > 60 ml/min (Cockcroft-Gault formula); Urine analysis results showing urinary protein (UPRO) < 2+ or 24-hour urinary protein < 1g;

   Cardiac function:
   * New York Heart Association (NYHA) class < 3;
   * Echocardiography showing left ventricular ejection fraction (LVEF) ≥ 50%;
9. For female subjects: should be surgically sterilized, postmenopausal patients, or agree to use at least one medically approved contraceptive method (such as intrauterine device [IUD], contraceptive pills, or condoms) during the study treatment period and for at least 6 months after the end of the study treatment. Serum or urine pregnancy test must be negative within 7 days before enrollment and must not be lactating. Male subjects should agree to use at least one medically approved contraceptive method (such as condoms, abstinence, etc.) during the study treatment period and for at least 6 months after the end of the study treatment;
10. Willing and able to comply with the trial and follow-up procedures.

Exclusion Criteria:

1. Patients with central nervous system metastases and/or carcinomatous meningitis. Patients who have undergone treatment for brain metastases may be considered for participation in this study provided that their condition has remained stable for at least 3 months, there is no evidence of disease progression on imaging performed within 4 weeks prior to the initiation of study treatment, all neurological symptoms have returned to baseline levels, there is no evidence of new or enlarging brain metastases, and there has been a discontinuation of radiation, surgery, or corticosteroid therapy for at least 28 days prior to the initiation of study treatment. This exception does not apply to carcinomatous meningitis, which should be excluded regardless of clinical stability.
2. Toxicities from prior anti-tumor therapy have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 0-1 (except for grade 2 alopecia).
3. Major surgery within 4 weeks prior to the start of study treatment and incomplete recovery.
4. Clinically significant pleural effusion or ascites requiring symptomatic treatment.
5. Receipt of attenuated live vaccines within 30 days prior to or anticipated during the study period.
6. Occurrence of a severe thromboembolic event or cerebrovascular accident within 1 year prior to study treatment initiation, such as deep vein thrombosis (excluding asymptomatic and non-interventional muscle venous thrombosis), pulmonary embolism, stroke, intracranial hemorrhage, myocardial infarction, except for asymptomatic and clinically non-interventional lacunar infarction.
7. Heart failure categorized as New York Heart Association (NYHA) class 3 or higher.
8. Presence of systemic diseases judged by the investigator to be unstable, including diabetes, hypertension, cirrhosis, interstitial pneumonia, obstructive lung disease, etc.
9. Active autoimmune disease requiring systemic therapy within 2 years prior to study treatment initiation (such as use of immunomodulatory drugs, corticosteroids, or immunosuppressants), with permitted alternative therapies (e.g., thyroid hormone, insulin, or physiological corticosteroid replacement therapy for renal or pituitary insufficiency).
10. Severe infection within 4 weeks prior to the first dose of study treatment (e.g., requiring intravenous administration of antibiotics, antifungals, or antiviral drugs), or occurrence of unexplained fever >38.5°C during the screening period or within 3 weeks prior to the first dose of study treatment.
11. Active autoimmune disease or immunodeficiency, or a history thereof, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, pituitary inflammation, vasculitis, nephritis, etc. Exceptions include patients with a history of autoimmune thyroiditis who receive thyroid hormone replacement therapy or patients with type 1 diabetes whose blood glucose is controlled with insulin therapy.
12. Active or poorly controlled severe infections, including:

    1. Human Immunodeficiency Virus (HIV) (positive for HIV1/2 antibodies);
    2. Active hepatitis B (positive for HBsAg or abnormal liver function with HBV DNA >2000IU/ml);
    3. Active hepatitis C (positive for HCV antibodies or HCV RNA ≥103 copies/ml with abnormal liver function);
    4. Active tuberculosis;
    5. Other uncontrollable active infections (CTCAE V5.0 > grade 2);
    6. Subjects who have received or plan to receive solid organ or hematopoietic stem cell transplantation during the study period (excluding corneal transplantation);
13. Subjects with a history of other malignant tumors within five years (except completely treated in situ cervical cancer, basal cell carcinoma, or squamous cell carcinoma of the skin);
14. Currently participating in interventional clinical research treatment or received other investigational drugs or investigational device therapy within 4 weeks prior to the first dose of study treatment. Subjects have not fully recovered from any intervention-induced toxicities and/or complications (i.e., ≤ grade 1 or returned to baseline, excluding fatigue or alopecia) before the first dose of study treatment;
15. Clear history of allergy or potential allergy or intolerance to investigational drugs and similar biological agents;
16. History of substance abuse involving psychotropic drugs and unable to abstain, or presence of psychiatric disorders;
17. Other conditions determined by the investigator to increase the risk associated with study participation or investigational drug, and according to the investigator's judgment, may render the patient unsuitable for study enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival，PFS | 21 or 28 days after the last dose
  To evaluate the efficacy of anti-tumor

SECONDARY OUTCOMES:
Overall survival，OS | 1 year after the last dose
  To evaluate the efficacy of anti-tumor
Objective response rate，ORR | 21 or 28 days after the last dose
  To evaluate the efficacy of anti-tumor
Disease Control Rate，DCR | 21 or 28 days after the last dose
  To evaluate the efficacy of anti-tumor
Duration of Response，DoR | 21 or 28 days after the last dose
  To evaluate the efficacy of anti-tumor
Safety: Hematologic and non-hematologic toxicity (NCI CTCAE v5.0) | rom the initiation of the first dose to 21 or 28 days after the last dose
  To identify the incidence of AE and SAE in clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Li, Dr., Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences